CLINICAL TRIAL: NCT02445417
Title: Brain Activity During Birth for Prediction of Newborns at Risk for Brain Injury
Status: Completed | Type: Observational
Sponsor: Sharp HealthCare (Other)
Collaborators: The Hartwell Foundation (Other)
Responsible Party: Principal Investigator, M J Harbert, Director of Neonatal Neurology, Sharp HealthCare
Other Study IDs: Transition
Record Dates: First submitted 2015-03-31; First posted 2015-05-15 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Encephalopathy; Asphyxia Newborns
Keywords: Perinatal depression
MeSH Terms: conditions — Brain Diseases; Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EES: Epidermal Electronic System
- Hydrogel Electrode: Hydrogel based EEG electrode

SUMMARY:
The purpose of this study is early identification of asphyxiated newborns through eeg starting in the delivery room.

DETAILED DESCRIPTION:
There is a need for a reliable detector of birth asphyxia so that newborns with birth asphyxia can have timely and accurate diagnosis to receive therapeutic hypothermia within 6 hrs of life, which has been shown to significantly reduce deaths and improve long term developmental outcomes.

This study is designed to record EEG during birth transition through the first 10 minutes of life.

ELIGIBILITY:
Inclusion Criteria: Term infants

* Signed Informed consent

Exclusion Criteria:

* Known congenital anomalies

Ages: 36 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term infants at delivery (37-44 weeks gestational age)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
EEG recorded | Birth to 10 minutes of life
  May be up to 60 minutes if applicable

SECONDARY OUTCOMES:
Skin irritation from EES or hydrogel electrodes | 60 minutes of life
  Redness, excoriation
Successful adhesion of EES to skin | 60 minutes of life
  Redness, excoriation

OTHER OUTCOMES:
Apgar scores | Birth to 10 minutes of life
  At 1, 5, 10, 15 and 20 minutes of life if done
Blowby oxygen at delivery | Birth to 10 minutes of life
Intubation at delivery | Birth to 10 minutes of life
  for meconium suctioning or ventilation purposes
Positive Pressure Ventilation | Birth to 10 minutes of life
  By bag and mask or endotracheal tube
Continuous Positive Airway Pressure | Birth to 10 minutes of life
Epinephrine administration | Birth to 10 minutes of life
Sodium bicarbonate administration | Birth to 10 minutes of life
Normal saline bolus administration | Birth to 10 minutes of life
Chest compressions | Birth to 10 minutes of life
Near-infrared spectroscopy measurement | Birth to 10 minutes of life. May extend to 60 minutes of life if applicable.
  Non-invasive brain tissue oximetry recording

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Harbert, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

REFERENCES:
- [Background] Raghuveer TS, Cox AJ. Neonatal resuscitation: an update. Am Fam Physician. 2011 Apr 15;83(8):911-8. PMID 21524031
- [Background] Perez A, Ritter S, Brotschi B, Werner H, Caflisch J, Martin E, Latal B. Long-term neurodevelopmental outcome with hypoxic-ischemic encephalopathy. J Pediatr. 2013 Aug;163(2):454-9. doi: 10.1016/j.jpeds.2013.02.003. Epub 2013 Mar 14. PMID 23498155
- [Background] Massaro AN, Tsuchida T, Kadom N, El-Dib M, Glass P, Baumgart S, Chang T. aEEG evolution during therapeutic hypothermia and prediction of NICU outcome in encephalopathic neonates. Neonatology. 2012;102(3):197-202. doi: 10.1159/000339570. Epub 2012 Jul 12. PMID 22796967
- [Background] Jacobs SE, Berg M, Hunt R, Tarnow-Mordi WO, Inder TE, Davis PG. Cooling for newborns with hypoxic ischaemic encephalopathy. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003311. doi: 10.1002/14651858.CD003311.pub3. PMID 23440789
- [Background] Shalak LF, Laptook AR, Velaphi SC, Perlman JM. Amplitude-integrated electroencephalography coupled with an early neurologic examination enhances prediction of term infants at risk for persistent encephalopathy. Pediatrics. 2003 Feb;111(2):351-7. doi: 10.1542/peds.111.2.351. PMID 12563063
- [Background] Kim DH, Lu N, Ma R, Kim YS, Kim RH, Wang S, Wu J, Won SM, Tao H, Islam A, Yu KJ, Kim TI, Chowdhury R, Ying M, Xu L, Li M, Chung HJ, Keum H, McCormick M, Liu P, Zhang YW, Omenetto FG, Huang Y, Coleman T, Rogers JA. Epidermal electronics. Science. 2011 Aug 12;333(6044):838-43. doi: 10.1126/science.1206157. PMID 21836009
- [Background] Pichler G, Avian A, Binder C, Zotter H, Schmolzer GM, Morris N, Muller W, Urlesberger B. aEEG and NIRS during transition and resuscitation after birth: promising additional tools; an observational study. Resuscitation. 2013 Jul;84(7):974-8. doi: 10.1016/j.resuscitation.2012.12.025. Epub 2013 Jan 8. PMID 23313424
- See also: cdc: Complications during pregnancy & birth are among leading causes of infant mortality — http://cdc.gov/nchs/data/hestat/prelimdeaths05/prelimdeaths05.htm.